CLINICAL TRIAL: NCT05031299
Title: Lifestyle-related Early Detection and Intervention for Older Adults & Elderly at Risk for Metabolic Syndrome: GATEKEEPER
Brief Title: Lifestyle-related Early Detection and Intervention for Older Adults & Elderly at Risk for Metabolic Syndrome
Acronym: GATEKEEPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harokopio University (Other)
Collaborators: CitiesNet (Unknown); University of Thessaly (Other); University of Patras (Other); BioAssist (Unknown); University of Ioannina (Other); Centre for Research & Technology Hellas (CERTH) (Unknown)
Responsible Party: Principal Investigator, Yannis Manios, Professor, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 488; 857223 (Other Grant/Funding Number: European Union Horizon 2020 research & innovation programme)
Record Dates: First submitted 2021-07-29; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; lifestyle intervention; prevention; digital tools; elderly; older adults
MeSH Terms: conditions — Metabolic Syndrome | interventions — Standard of Care; Self-Management; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: The present study is a cluster-randomized lifestyle intervention aimed at primary and secondary prevention of MetS, including three study arms: standard care (control group), standard care plus lifestyle application (intervention group 1) and standard care plus lifestyle application and wearables and devices (intervention group 2). It is conducted with older adults and elderly (aged ≥55 years old) living at home and at risk for MetS, as well as their carers. The total duration of the intervention for each participant will be 3 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Standard care) (Active Comparator): Participants in the control group will receive only the standard care as provided by the local and national healthcare system as well as one face-to-face counselling session for lifestyle modification to improve their risk factors for 3 months.
  Interventions: Behavioral: Standard care
- Intervention group 1 (Application) (Experimental): Participants will will be additionally provided with a health-promotion application for self-management for 3 months.
  Interventions: Behavioral: Health-promotion application for self-management
- Intervention group 2 (Devices) (Experimental): Participants will be additionally provided with wearables and devices for 3 months including:
  * A weighing scale (assessing also body composition) device
  * A smartwatch/wristband to assess physical activity but also sleep pattern.
  Interventions: Device: Wearables and devices

INTERVENTIONS:
Behavioral: Standard care — Participants will receive only the standard care as provided by the local and national healthcare system as well as one face-to-face counselling session for lifestyle modification to improve their risk factors.
  Arms: Control group (Standard care)
Behavioral: Health-promotion application for self-management — Participants will be provided with a health-promotion application for self-management for 3 months, additionally to the standard care.
  Arms: Intervention group 1 (Application)
Device: Wearables and devices — Participants will be provided with wearables and devices, including a weighing scale (assessing also body composition) device and a smartwatch/wristband to assess physical activity but also sleep pattern, for 3 months, additionally to the standard care and the Health-promotion application.
  Arms: Intervention group 2 (Devices)

SUMMARY:
In GATEKEEPER intervention, Big Data Analytics techniques will be exploited to address risk stratification and early detection, based on lifestyles analysis including: pattern recognition for the improvement of public health surveillance and for the early detection of chronic conditions; data mining for inductive reasoning and exploratory data analysis; Cluster Analysis for identifying high-risk groups among elder citizens. In the above cases timely intervention is provided by through AI-based, digital coaches, structured conversations, consultation and education. The main target group (N=960) is older adults and elderly citizens with risk factors for MetS and their carers. Therefore, the GATEKEEPER intervention aims at primary (avoid occurrence of disease) and secondary (early detection and management) prevention of the ageing population at risk for MetS.

DETAILED DESCRIPTION:
Over 1.5 billion people worldwide are affected by Metabolic Syndrome (MetS) - a cluster of conditions reflecting behavioural risk factors typical of modern lifestyle (excessive food intake, low physical activity, etc) - with a huge socioeconomic impact and a total estimated cost of trillions of euros.

Early prevention measures especially for elderly at high risk of chronic conditions, such as prediabetics or obese, include structured lifestyle change programs that help people achieve and sustain changes in dietary and physical activity habits.

It is well established that MetS prevalence, as well as its individual components (high blood pressure, high glucose, central adiposity) increase with age. Notably, MetS percentages in the age group 50-55 years old and older is almost 2-3 times higher than in the younger age groups, probably due to a life time accumulation of adversities including overnutrition, a sedentary lifestyle, obesity and dyslipidemia, changes in the hormones, untreated hypertension, changes of the functioning of beta cells and other environmental and physiological factors.

Therefore, it is important to target not only elderly citizens, but rather older adults aged ≥55 years old as the optimum target group for a MetS prevention intervention.

In GATEKEEPER intervention, Big Data Analytics techniques will be exploited to address risk stratification and early detection, based on lifestyles analysis including: pattern recognition for the improvement of public health surveillance and for the early detection of chronic conditions; data mining for inductive reasoning and exploratory data analysis; Cluster Analysis for identifying high-risk groups among elder citizens. In the above cases timely intervention is provided by through AI-based, digital coaches, structured conversations, consultation and education. The main target group (N=960) is older adults and elderly citizens with risk factors for MetS and their carers. Therefore, the GATEKEEPER intervention aims at primary (avoid occurrence of disease) and secondary (early detection and management) prevention of the ageing population at risk for MetS.

960 older adults and elderly citizens (aged >=55 years old) with risk factors for MetS as well as their carers (n=40) will be recruited and will be randomized to either: i) the intervention group 1 (n=320), who will be provided with the standard care plus a lifestyle application to promote self-management, increase health literacy and awareness through a digital coach, ii) the intervention group 2 (n=320), who will be provided with the standard care, the lifestyle application and additionally digital tools and wearables, such as a smart tracker and weight scale, or iii) the control group (n=320), who will only receive standard care, as provided by the local and national healthcare system as well as one face-to-face counselling session for lifestyle modification to improve their risk factors.

The participants will be followed up for a total duration of 3 months, when they will be re-evaluated to assess whether their risk factors were improved through the lifestyle intervention.

The users will be recruited at local community centres, such as the "Open Day Elderly Centres", health centres, private offices of health care professionals, hospitals etc. upon written informed consent form.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥55 years old
* Having any of the following risk factors for MetS:

  * waist circumference >94 cm for men and >80 cm for women
  * Triglycerides (TG) ≥150 mg/dL
  * High-density lipoprotein cholesterol (HDL-C) <40 mg/dL for men and <50 mg/dL for women
  * Fasting glucose ≥100 mg/dL
  * Blood pressure ≥130 /≥85 mm Hg
* Living at home (either alone or with relatives)
* Informed consent form provided

Exclusion Criteria:

* Having severe hearing or vision problems or any other acute or chronic condition that would limit the ability of the user to participate in the study
* Having dementia or cognitive impairment
* Being institutionalised
* Participation in another research project

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Waist circumference (cm) from baseline to 3 months | baseline and monthly until 3-month follow-up
  Participants' waist circumference will be measured in triplicates (in cm) at baseline and at the 3rd month follow-up visit.

SECONDARY OUTCOMES:
Changes in body mass index (kg/m2) from baseline to 3 months | baseline and monthly until 3-month follow-up
  Participants' BMI will be measured in triplicates (in kg/m2) at baseline and at the 3rd month follow-up visit.
Changes in percentage of body fat from baseline to 3 months | baseline and monthly until 3-month follow-up
  Participants' percentage of body fat will be measured at baseline and at the 3rd month follow-up visit.
Patient-reported outcome measures (PROMs) | baseline and 3 months
  Patient-reported outcome measures (PROMs), including satisfaction of the intervention at baseline and at the 3rd month follow-up visit. Satisfaction of the intervention will be measured via the UTAUT questionnaire [Liu D et al. 2019] or other validated questionnaire.
Changes in Diet quality on FFQ and healthy diet score from baseline to 3 months | baseline and 3 months
  Diet quality will be assessed via the food-frequency questionnaire (FFQ) and the healthy diet score developed and validated in the EU-funded Feel4Diabetes-study (www.feel4diabetes-study.eu) or other validated questionnaires at baseline and at the 3rd month follow-up visit.
Changes in Quality of life on EQ5D (Generic HRQL) from baseline to 3 months | baseline and 3 months
  Quality of life will be assessed via the EQ5D (Generic HRQL) [Konerding U et al. 2014] at baseline and at the 3rd month follow-up visit.
Changes in Physical activity on validated questionnaires from baseline to 3 months | baseline and 3 months
  Physical activity will be assessed via validated questionnaires at baseline and at the 3rd month follow-up visit.
Changes in sedentary time on validated questionnaires from baseline to 3 months | baseline and 3 months
  Sedentary time will be assessed via validated questionnaires at baseline and at the 3rd month follow-up visit.
Changes in Sleep duration/quality on Athens Insomnia Scale questionnaire from baseline to 3 months | baseline and 3 months
  Sleep duration and sleep quality will be assessed via the Athens Insomnia Scale questionnaire [Soldatos CR et al. 2000] or other validated questionnaires at baseline and at the 3rd month follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Odysseas Androutsos, PhD, Principal Investigator — University of Thessaly
Locations (2):
- Greece (2):
  - Harokopio University of Athens, Kallithea, Attica
  - University of Thessaly, Trikala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimmet P, M M Alberti KG, Serrano Rios M. [A new international diabetes federation worldwide definition of the metabolic syndrome: the rationale and the results]. Rev Esp Cardiol. 2005 Dec;58(12):1371-6. No abstract available. Spanish. PMID 16371194
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Saklayen MG. The Global Epidemic of the Metabolic Syndrome. Curr Hypertens Rep. 2018 Feb 26;20(2):12. doi: 10.1007/s11906-018-0812-z. PMID 29480368
- [Background] Lesjak V, Stanojevic-Jerkovic O. Physical Activity, Sedentary Behavior and Substance Use among Adolescents in Slovenian Urban Area. Zdr Varst. 2015 Jun 9;54(3):168-74. doi: 10.1515/sjph-2015-0024. eCollection 2015 Sep. PMID 27646724
- [Background] Scuteri A, Laurent S, Cucca F, Cockcroft J, Cunha PG, Manas LR, Mattace Raso FU, Muiesan ML, Ryliskyte L, Rietzschel E, Strait J, Vlachopoulos C, Volzke H, Lakatta EG, Nilsson PM; Metabolic Syndrome and Arteries Research (MARE) Consortium. Metabolic syndrome across Europe: different clusters of risk factors. Eur J Prev Cardiol. 2015 Apr;22(4):486-91. doi: 10.1177/2047487314525529. Epub 2014 Mar 19. PMID 24647805
- [Background] Devers MC, Campbell S, Simmons D. Influence of age on the prevalence and components of the metabolic syndrome and the association with cardiovascular disease. BMJ Open Diabetes Res Care. 2016 Apr 25;4(1):e000195. doi: 10.1136/bmjdrc-2016-000195. eCollection 2016. PMID 27158519
- [Background] Kraja AT, Borecki IB, North K, Tang W, Myers RH, Hopkins PN, Arnett D, Corbett J, Adelman A, Province MA. Longitudinal and age trends of metabolic syndrome and its risk factors: the Family Heart Study. Nutr Metab (Lond). 2006 Dec 5;3:41. doi: 10.1186/1743-7075-3-41. PMID 17147796
- [Background] Athyros VG, Ganotakis ES, Bathianaki M, Monedas I, Goudevenos IA, Papageorgiou AA, Papathanasiou A, Kakafika AI, Mikhailidis DP, Elisaf M; MetS-Greece Collaborative Group. Awareness, treatment and control of the metabolic syndrome and its components: a multicentre Greek study. Hellenic J Cardiol. 2005 Nov-Dec;46(6):380-6. PMID 16422124
- [Background] Park MJ, Kim HS. Evaluation of mobile phone and Internet intervention on waist circumference and blood pressure in post-menopausal women with abdominal obesity. Int J Med Inform. 2012 Jun;81(6):388-94. doi: 10.1016/j.ijmedinf.2011.12.011. Epub 2012 Jan 21. PMID 22265810
- [Background] Konerding U, Elkhuizen SG, Faubel R, Forte P, Malmstrom T, Pavi E, Janssen MF. The validity of the EQ-5D-3L items: an investigation with type 2 diabetes patients from six European countries. Health Qual Life Outcomes. 2014 Dec 5;12:181. doi: 10.1186/s12955-014-0181-5. PMID 25479769
- [Background] Kokaliari ED, Roy AW. Validation of the Greek translation of the multicultural quality of life index (MQLI-gr). Health Qual Life Outcomes. 2020 Jun 15;18(1):183. doi: 10.1186/s12955-020-01426-9. PMID 32539776
- [Background] Liu D, Maimaitijiang R, Gu J, Zhong S, Zhou M, Wu Z, Luo A, Lu C, Hao Y. Using the Unified Theory of Acceptance and Use of Technology (UTAUT) to Investigate the Intention to Use Physical Activity Apps: Cross-Sectional Survey. JMIR Mhealth Uhealth. 2019 Aug 22;7(9):e13127. doi: 10.2196/13127. PMID 31507269
- [Background] Soldatos CR, Dikeos DG, Paparrigopoulos TJ. Athens Insomnia Scale: validation of an instrument based on ICD-10 criteria. J Psychosom Res. 2000 Jun;48(6):555-60. doi: 10.1016/s0022-3999(00)00095-7. PMID 11033374